CLINICAL TRIAL: NCT06387745
Title: Use of Ultrasound Tools to Refer Patients at Risk of Chronic Liver Disease to the Hepatology Consultation (US-REFERRAL)
Brief Title: Referral of Patients to Hepatology With Hepatoscope
Acronym: US-REFERRAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: E-Scopics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: US-REFERRAL
Record Dates: First submitted 2024-04-17; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Investigational Arm (Experimental): Single arm study protocol
  Interventions: Device: Hepatoscope

INTERVENTIONS:
Device: Hepatoscope — The Hepatoscope is a non-invasive external ultrasound imaging device, intended for general purpose pulse echo ultrasound imaging, and soft tissue elasticity imaging of the human body. In addition, the Hepatoscope provides measurements of shear wave speed and tissue stiffness, ultrasound beam attenuation and estimates of speed of sound, in internal structures of the body.

SUMMARY:
Patients identified as being at risk of liver fibrosis because of a positive Fibrosis-4 (FIB-4) test in the primary care setting will be offered be enrolled in the trial and to undergo an Hepatoscope exam (external non-invasive ultrasound imaging exam) to screen for liver fibrosis (with stiffness measurements) and/or steatosis (with ultrasound parameters related to fatty liver). All patients presenting with a liver stiffness value of at least 6.5 kilopascal (kPa) will be referred to the tertiary hepatology consultations for further assessment. Hepatoscope measurements will be compared to the standard of care for these patients, as defined at the tertiary hepatology center.

DETAILED DESCRIPTION:
Chronic liver diseases (CLD) remain asymptomatic for a long time, until they become decompensated (cirrhosis) or lead to liver cancer. CLD all have a very similar natural history: over several years, or even tens of years, liver fibrosis develops progressively, which leads to cirrhosis and the related risks of complications of cirrhosis, including portal hypertension, liver failure, of even liver cancer.

In the absence of complications, liver fibrosis and cirrhosis remain completely symptomatic. For this reason, several methods for the non-invasive assessment of liver fibrosis have been developed over the last 20 years, with the objective to screen for liver fibrosis in it early stage so as to manage the patient and potentially prevent to development of complications. There are 2 groups of such noninvasive methods: blood-based tests and methods that measure the liver stiffness, which is directly correlated to liver fibrosis severity.

There are simple blood tests such as the FIB-4 and others can be more complex like FibroTest.

The FIB-4 test, which takes into account 4 parameters easily available (age, platelets, and 2 liver enzymes, AST and ALT), is very useful in the general population because of its high negative predictive value. However, it is mainly used for the diagnosis of liver fibrosis in the context of chronic viral hepatitis.

The measurement of liver stiffness is currently available on a hepatology-dedicated device, the FibroScan, or on high-end ultrasound imaging systems that are available in radiology centers. This measurement of liver stiffness has demonstrated excellent performances for the diagnosis of cirrhosis and a good performance for the assessment of liver fibrosis severity at earlier stages. However, in clinical practice, this method is not widely available nor accessible (cost of equipment of limited to radiology centers).

For the diagnosis of liver steatosis (excess of fat accumulation in the liver), which can also lead to liver fibrosis, cirrhosis and its complications, the Gold Standard exam that can quantify the extent of fat in the liver is Magnetic Resonance Imaging derived Proton Density Fat Fraction (MRI PDFF), but its use in routine is extremely limited due to the lack of MRI equipment, their cost, and the cost of MRI exams. Liver steatosis can be assessed with ultrasound imaging systems (in radiology) and also with FibroScan, although the interpretation of exam results remains variable.

In primary care, in diabetology-endocrinology and in the hepatology practice, it is now known that the screening of chronic liver diseases at their early stages is of paramount importance for a proper management of patients. New simple, available and affordable tools are urgently needed to cover the territory and assess patients at risk where they are, at the point of care, during consultations.

This clinical trial will assess the performance of an ultra-portable, point-of-care ultrasound device for the assessment of liver fibrosis and steatosis in the primary care setting, to optimize referral of patients to the tertiary hepatology consultation for further specialist investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any of the following

  * Elevated liver enzymes (AST, ALT, Gamma-GT, AP)
  * Type 2 diabetes
  * Elements of metabolic syndrome
* Patients who consent in written to participate in the Clinical Investigation after being orally informed on the objectives and methods of the Clinical Investigation

Exclusion Criteria:

* Patients with active implants such as pacemakers, defibrillators, pumps, etc.
* Patients presenting wounds at the location where the Hepatoscope probe shall be placed on patients' skin,
* Pregnant and breastfeeding women,
* People deprived of their freedom rights.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value for significant fibrosis | at study completion: 12 months
  Estimation of Positive Predictive Value in percentage with 95% confidence interval for estimation of significant fibrosis.

SECONDARY OUTCOMES:
Correlation of stiffness measurements | at study completion: 12 months
  Liver stiffness measurements performed with the device subject of the research and competitor device will be compared by analysis of correlation. The analysis outcome will be the R² coefficient and its p value.
Concordance of stiffness measurements | at study completion: 12 months
  Liver stiffness measurements performed with the device subject of the research and competitor device will be compared by analysis of concordance. The analysis outcome will be the Concordance Correlation Coefficients (CCC) and 95% confidence intervals.
Diagnostic performance of liver stiffness measurements | at study completion: 12 months
  Area under the receiver operating characteristic (ROC) curve will be used an a general assessment of diagnostic performance against dichotomized population according to referral outcome. Diagnostic estimators in the studied population will be derived from the ROC analysis: sensitivity, specificity, positive and negative predictive values.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Vonghia, MD, PhD, Principal Investigator — University Hospital, Antwerp

IPD SHARING:
Plan to Share IPD: No